CLINICAL TRIAL: NCT01230736
Title: Assessing the Safety and Efficacy of Changing to DuoTrav® (Travoprost 0.004%/Timolol 0.5% Fixed Combination) as Replacement Therapy in Patients Uncontrolled on Bimatoprost 0.03%/Timolol 0.5% Therapy (Fixed or Unfixed)
Brief Title: Safety and Efficacy of Changing to DuoTrav From Prior Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-10-243
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2012-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav (Experimental): One drop in study eye(s) once daily for 8 weeks
  Interventions: Drug: Travoprost 0.004%/Timolol 0.5% Fixed Combination eye drops solution (Duotrav®)

INTERVENTIONS:
Drug: Travoprost 0.004%/Timolol 0.5% Fixed Combination eye drops solution (Duotrav®) — One drop in study eye(s) once daily for 8 weeks
  Other Names: DuoTrav®

SUMMARY:
The purpose of this study to assess the safety and efficacy of changing to DuoTrav® from prior bimatoprost 0.03%/timolol 0.5% (used concomitantly or in a fixed combination) pharmacotherapy in uncontrolled patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in both eyes.
* Must have an IOP of between 19 to 35 millimeters mercury (mmHg) (at any time of the day) in at least one eye (which would be designated as the study eye).
* Must be willing to discontinue the use of all other ocular hypotensive medication(s) prior to receiving the study medication for the entire course of the study.
* Women who are pregnant or lactating.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of DuoTrav® that is deemed clinically significant in the opinion of the Principal Investigator.
* Corneal dystrophies in either eye.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Bronchial asthma or a history of bronchial asthma, bronchial hyper-reactivity, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* History of severe allergic rhinitis.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) at 8 weeks from prior therapy (baseline) | 8 weeks
  Goldmann applanation tonometry will be performed at the baseline visit and 8-week visit to record intraocular pressure (IOP). The difference between the two readings will be recorded as the change in IOP. IOP will be recorded in mmHg.

SECONDARY OUTCOMES:
Percentage of subjects who reach target IOP (≤18 mmHg) | 8 weeks
  Goldmann applanation tonometry will be performed at the 8-week visit to record intraocular pressure. Percentage of patients who reach target IOP will be calculated by comparing patients with IOP ≤18 mmHg to the overall study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Schweinfurt, Germany

REFERENCES:
- [Result] Scherzer ML, Liehneova I, Negrete FJ, Schnober D. Travoprost 0.004%/timolol 0.5% fixed combination in patients transitioning from fixed or unfixed bimatoprost 0.03%/timolol 0.5%. Adv Ther. 2011 Aug;28(8):661-70. doi: 10.1007/s12325-011-0043-z. Epub 2011 Jul 15. PMID 21773673